CLINICAL TRIAL: NCT01684722
Title: Vitamin D and Omega-3 Trial to Prevent and Treat Diabetic Kidney Disease
Acronym: VITAL-DKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Brigham and Women's Hospital (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ian deBoer, Associate Professor, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 39113; R01DK088762 (NIH)
Record Dates: First submitted 2012-09-06; First posted 2012-09-13 (Estimated); Results first posted 2020-06-26 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Diabetes
Keywords: vitamin D3; omega-3 fatty acids; fish oil; diabetes; kidney disease; albuminuria; urine albumin excretion; glomerular filtration rate; diabetic kidney disease
MeSH Terms: conditions — Diabetes Mellitus; Kidney Diseases; Albuminuria; Diabetic Nephropathies | interventions — Vitamin D; Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin D + fish oil (Active Comparator): Vitamin D and omega-3 fatty acids (fish oil)
  Interventions: Dietary Supplement: Vitamin D; Drug: Omega-3 fatty acids (fish oil)
- Vitamin D + fish oil placebo (Active Comparator): Vitamin D and fish oil placebo
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: Fish oil placebo
- Vitamin D placebo + fish oil (Active Comparator): Vitamin D placebo and omega-3 fatty acids (fish oil)
  Interventions: Drug: Omega-3 fatty acids (fish oil); Dietary Supplement: Vitamin D placebo
- Vitamin D placebo + fish oil placebo (Placebo Comparator): Vitamin D placebo and fish oil placebo
  Interventions: Dietary Supplement: Vitamin D placebo; Dietary Supplement: Fish oil placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D3 (cholecalciferol), 2000 IU per day.
  Arms: Vitamin D + fish oil; Vitamin D + fish oil placebo
Drug: Omega-3 fatty acids (fish oil) — Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Arms: Vitamin D + fish oil; Vitamin D placebo + fish oil
Dietary Supplement: Vitamin D placebo — Vitamin D3 placebo
  Arms: Vitamin D placebo + fish oil; Vitamin D placebo + fish oil placebo
Dietary Supplement: Fish oil placebo — Fish oil placebo
  Arms: Vitamin D + fish oil placebo; Vitamin D placebo + fish oil placebo

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259) is a randomized clinical trial in 20,000 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or fish oil (1 gram of omega-3 fatty acids) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. This ancillary study is being conducted among participants in VITAL with a history of diabetes and will examine whether vitamin D or fish oil prevents the development and progression of diabetic kidney disease.

DETAILED DESCRIPTION:
This ancillary study to the VITamin D and OmegA-3 TriaL (VITAL) will test whether vitamin D3, omega-3 fatty acids, or both prevent the development and progression of diabetic kidney disease (DKD). Persons with diabetes are at high risk of kidney disease. In 2005-2008, the prevalence of DKD among people with type 2 diabetes in the United States was 34.5%. Moreover, from 1988-1994 to 2005-2008, the prevalence of DKD in the United States grew 34% to 6.9 million people. DKD is both the leading cause of end stage renal disease in the developed world and a potent amplifier of cardiovascular disease risk.

Vitamin D and omega-3 fatty acids are promising interventions for DKD prevention and treatment, based on results of animal-experimental models and early human studies. Because these interventions are relatively safe, inexpensive, and widely available, they may offer opportunity to substantially reduce the burden of DKD in large populations. This VITAL ancillary study will test whether vitamin D3 and/or omega-3 fatty acids prevent progression of albuminuria and loss of glomerular filtration rate, two complementary manifestations of DKD, over 3 years of treatment.

In VITAL, 20,000 participants will be randomly assigned in a 2x2 factorial design to vitamin D3 (cholecalciferol) 2000 IU daily versus placebo, and to eicosapentaenoic acid 465 mg plus docosahexaenoic acid 375 mg daily versus placebo, and followed for a mean of 5 years to assess effects on cardiovascular disease and cancer events. This ancillary study will identify and recruit a sub-cohort of VITAL participants with diabetes at baseline and ascertain effects of study interventions on albuminuria and glomerular filtration rate in this group. First morning voids will be collected at baseline and year 3 for measurement of urine albumin-creatinine ratio. Blood samples will be collected simultaneously for measurement of estimated glomerular filtration rate (using serum creatinine and cystatin C) and other relevant biomarkers. This VITAL ancillary study is designed to determine whether vitamin D3 and/or omega-3 fatty acids have causal and clinically relevant effects on the development and progression of DKD.

ELIGIBILITY:
Inclusion Criteria: Participants in VITAL (NCT 01169259) with a self-reported physician diagnosis of diabetes are eligible to participate in this ancillary study.

Exclusion Criteria:

* Type 1 diabetes
* Diabetes only during pregnancy
* Known cause of kidney disease other than diabetes
* History of kidney transplantation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1312 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian H de Boer, MD, MS, Principal Investigator — University of Washington
Locations (1):
- Brigham Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Best CM, Zelnick LR, Thummel KE, Hsu S, Limonte C, Thadhani R, Sesso HD, Manson JE, Buring JE, Mora S, Lee IM, Cook NR, Friedenberg G, Luttmann-Gibson H, de Boer IH, Hoofnagle AN. Serum Vitamin D: Correlates of Baseline Concentration and Response to Supplementation in VITAL-DKD. J Clin Endocrinol Metab. 2022 Jan 18;107(2):525-537. doi: 10.1210/clinem/dgab693. PMID 34543425
- [Derived] Limonte CP, Zelnick LR, Ruzinski J, Hoofnagle AN, Thadhani R, Melamed ML, Lee IM, Buring JE, Sesso HD, Manson JE, de Boer IH. Effects of long-term vitamin D and n-3 fatty acid supplementation on inflammatory and cardiac biomarkers in patients with type 2 diabetes: secondary analyses from a randomised controlled trial. Diabetologia. 2021 Feb;64(2):437-447. doi: 10.1007/s00125-020-05300-7. Epub 2020 Oct 24. PMID 33098434
- [Derived] de Boer IH, Zelnick LR, Ruzinski J, Friedenberg G, Duszlak J, Bubes VY, Hoofnagle AN, Thadhani R, Glynn RJ, Buring JE, Sesso HD, Manson JE. Effect of Vitamin D and Omega-3 Fatty Acid Supplementation on Kidney Function in Patients With Type 2 Diabetes: A Randomized Clinical Trial. JAMA. 2019 Nov 19;322(19):1899-1909. doi: 10.1001/jama.2019.17380. PMID 31703120
- See also: Vitamin D and Omega-3 Trial study website — http://www.vitalstudy.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D + Fish Oil Placebo | Vitamin D Placebo + Fish Oil | Vitamin D Placebo + Fish Oil Placebo | Vitamin D + Fish Oil
Started | 333 | 289 | 320 | 370
Completed | 236 | 212 | 226 | 260
Not Completed | 97 | 77 | 94 | 110
Not completed — Lost to Follow-up | 78 | 56 | 75 | 89
Not completed — Death | 19 | 21 | 19 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D + Fish Oil Placebo | Vitamin D Placebo + Fish Oil | Vitamin D Placebo + Fish Oil Placebo | Vitamin D + Fish Oil | Total
Number analyzed (Participants) | 333 | 289 | 320 | 370 | 1312
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (6.7) | 68.2 (6.7) | 67.5 (6.9) | 67.4 (7.3) | 67.6 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 131 | 151 | 184 | 609
  Male | 190 | 158 | 169 | 186 | 703
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic white | 211 | 199 | 207 | 240 | 857
  Non-Hispanic black | 75 | 59 | 71 | 73 | 278
  Hispanic | 21 | 16 | 18 | 20 | 75
  Asian/Pacific Islander | 8 | 7 | 7 | 13 | 35
  American Indian/Alaska Natuve | 4 | 1 | 2 | 6 | 13
  Other | 8 | 2 | 9 | 9 | 28
  Not available | 6 | 5 | 6 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Estimated Glomerular Filtration Rate
Description: GFR estimated from serum creatinine and cystatin C
Time Frame: baseline to 5 years
Population: Outcomes analyzed according to factorial assignments, without evidence of treatment interaction.
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73m2
Groups:
- Vitamin D: Vitamin D 2000IU daily
- Vitamin D Placebo; Fish Oil Placebo: Matching placebo daily
- Fish Oil: Fish oil one capsule daily
Arm/Group | Vitamin D | Vitamin D Placebo | Fish Oil | Fish Oil Placebo
Number analyzed (Participants) | 703 | 609 | 659 | 653
mL/min/1.73m2 | -12.3 [-13.4 to -11.2] | -13.1 [-14.2 to -11.9] | -12.2 [-13.3 to -11.1] | -13.1 [-14.2 to -12.0]
Statistical Analysis 1: Comparison: Vitamin D vs Vitamin D Placebo; Test type: Superiority; p = 0.25, Mixed Models Analysis; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-0.7 to 2.5]
Statistical Analysis 2: Comparison: Fish Oil vs Fish Oil Placebo; Test type: Superiority; p = 0.27, Mixed Models Analysis; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-0.7 to 2.6]

2. Secondary Outcome: Change in Urine Albumin Excretion
Description: Change in urine albumin-creatinine ratio.
Time Frame: baseline to 5 years
Population: Outcomes analyzed according to factorial assignments, without evidence of treatment interaction.
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean ratio
Arm/Group | Vitamin D | Vitamin D Placebo | Fish Oil | Fish Oil Placebo
Number analyzed (Participants) | 703 | 609 | 659 | 653
geometric mean ratio | 2.97 [2.66 to 3.32] | 3.02 [2.70 to 3.38] | 2.94 [2.62 to 3.30] | 3.05 [2.74 to 3.40]
Statistical Analysis 1: Comparison: Vitamin D vs Vitamin D Placebo; Test type: Superiority; p = 0.90, Mixed Models Analysis; Ratio of change from baseline, active to = 0.99, 95% CI 2-sided [0.84 to 1.17]
Statistical Analysis 2: Comparison: Fish Oil vs Fish Oil Placebo; Test type: Superiority; p = 0.64, Mixed Models Analysis; Ratio of change from baseline, active to = 0.96, 95% CI 2-sided [0.81 to 1.14]

3. Secondary Outcome: Change in C-reactive Protein
Description: Changes in serum concentrations in CRP
Time Frame: baseline to 5 years
Measure: Geometric Mean (Standard Deviation); unit: mg/L
Groups:
- Vitamin D Placebo: Vitamin D placebo group
- Fish Oil: Omega-3 fatty acids (fish oil): Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
- Fish Oil Placebo: Fish oil placebo group
Arm/Group | Vitamin D | Vitamin D Placebo | Fish Oil | Fish Oil Placebo
Number analyzed (Participants) | 703 | 609 | 659 | 653
mg/L | 0.93 (2.71) | 1.03 (3.03) | 0.90 (2.82) | 1.05 (2.89)

4. Secondary Outcome: Change in Interleukin-6
Description: Changes in serum concentrations in IL-6
Time Frame: baseline to 5 years
Measure: Geometric Mean (Standard Deviation); unit: pg/ml
Arm/Group | Vitamin D | Vitamin D Placebo | Fish Oil | Fish Oil Placebo
Number analyzed (Participants) | 703 | 609 | 659 | 653
pg/ml | 1.04 (4.48) | 1.09 (4.44) | 1.10 (4.33) | 1.02 (4.60)

5. Secondary Outcome: Change in NT-proBNP
Description: Changes in serum concentrations in NT-proBNP
Time Frame: baseline to 5 years
Population: 2x2 factorial design
Measure: Geometric Mean (Standard Deviation); unit: ng/l
Arm/Group | Vitamin D | Vitamin D Placebo | Fish Oil | Fish Oil Placebo
Number analyzed (Participants) | 703 | 609 | 659 | 653
ng/l | 1.72 (3.24) | 1.38 (3.02) | 1.56 (3.07) | 1.54 (3.24)

ADVERSE EVENTS:
Time Frame: Up to five years
Description: Only monitored safety conditions are reported.
Groups:
- Vitamin D + Fish Oil Placebo: Vitamin D and fish oil placebo Vitamin D: Vitamin D3 (cholecalciferol), 2000 IU per day. Fish oil placebo: Fish oil placebo
- Vitamin D Placebo + Fish Oil: Vitamin D placebo and omega-3 fatty acids (fish oil) Omega-3 fatty acids (fish oil): Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Vitamin D placebo: Vitamin D3 placebo
- Vitamin D Placebo + Fish Oil Placebo: Vitamin D placebo and fish oil placebo Vitamin D placebo: Vitamin D3 placebo Fish oil placebo: Fish oil placebo
- Vitamin D + Fish Oil: Vitamin D and omega-3 fatty acids (fish oil) Vitamin D: Vitamin D3 (cholecalciferol), 2000 IU per day. Omega-3 fatty acids (fish oil): Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
Arm/Group | Vitamin D + Fish Oil Placebo | Vitamin D Placebo + Fish Oil | Vitamin D Placebo + Fish Oil Placebo | Vitamin D + Fish Oil
All-Cause Mortality (participants affected / at risk) | 19/333 | 21/289 | 19/320 | 21/370
Serious Adverse Events (participants affected / at risk) | 45/333 | 59/289 | 45/320 | 44/370
Other Adverse Events (participants affected / at risk) | 134/333 | 135/289 | 133/320 | 136/370
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D + Fish Oil Placebo (N=333) | Vitamin D Placebo + Fish Oil (N=289) | Vitamin D Placebo + Fish Oil Placebo (N=320) | Vitamin D + Fish Oil (N=370)
Malignant cancer (General disorders) | 21 | 24 | 17 | 17
Cancer death (General disorders) | 6 | 5 | 5 | 2
Malignant breast cancer (General disorders) | 2 | 1 | 3 | 2
Malignant prostate cancer (General disorders) | 3 | 4 | 4 | 4
Malignant colorectal cancer (General disorders) | 3 | 1 | 1 | 0
Major CVD events (Cardiac disorders) | 15 | 13 | 18 | 16
Myocardial infarction (Cardiac disorders) | 6 | 6 | 8 | 6
Stroke (General disorders) | 8 | 5 | 4 | 6
Cardiovascular death (Cardiac disorders) | 4 | 5 | 7 | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D + Fish Oil Placebo (N=333) | Vitamin D Placebo + Fish Oil (N=289) | Vitamin D Placebo + Fish Oil Placebo (N=320) | Vitamin D + Fish Oil (N=370)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3) | 8 (8) | 2 (2) | 6 (6)
Kidney stones (Renal and urinary disorders) | 13 (13) | 12 (12) | 14 (14) | 19 (19)
Parathyroid condition (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Gastrointestinal bleeding (Gastrointestinal disorders) | 9 (9) | 18 (18) | 8 (8) | 10 (10)
Blood in urine (Renal and urinary disorders) | 30 (30) | 32 (32) | 29 (29) | 25 (25)
Easy bruising (Blood and lymphatic system disorders) | 98 (98) | 91 (91) | 97 (97) | 99 (99)
Frequent nosebleeds (Blood and lymphatic system disorders) | 12 (12) | 13 (13) | 17 (17) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2010-06-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT01684722/Prot_SAP_000.pdf
  • Informed Consent Form (2010-12-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT01684722/ICF_001.pdf